CLINICAL TRIAL: NCT06693349
Title: Evaluation of Platelet-rich Fibrin for Revascularization of Im-mature Permanent Teeth Versus Standard Apexification: a 12-month Clinical Follow-up Study
Brief Title: Evaluation of Platelet-rich Fibrin for Revascularization of Immature Permanent Teeth Versus Standard Apexification
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mohammed Nasser Alhajj (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Sponsor-Investigator, Mohammed Nasser Alhajj, Assistant Professor Dr. Mohammed Nasser Alhajj, Thamar University
Organization: Thamar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11111218
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: To Evaluate the Clinical and Radiographic Effect of Platelet-rich Fibrin in Treatment of Necrotic Permanent Teeth with Open Apices
Keywords: platelet-rich fibrin, revascularization, apexification

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Contaminated immature permanent teeth (Active Comparator): treatment of contaminated immature permanent teeth through either revascularization or apexification procedures
  Interventions: Drug: the effect of platelet-rich fibrin in treatment of contaminated and uncontaminated immature permanent teeth; Drug: the effect of apexification in treatment of contaminated and uncontaminated immature permanent teeth
- uncontaminated immature permanent teeth (Active Comparator): treatment of uncontaminated immature permanent teeth through either revascularization or apexification procedures
  Interventions: Drug: the effect of platelet-rich fibrin in treatment of contaminated and uncontaminated immature permanent teeth; Drug: the effect of apexification in treatment of contaminated and uncontaminated immature permanent teeth

INTERVENTIONS:
Drug: the effect of platelet-rich fibrin in treatment of contaminated and uncontaminated immature permanent teeth — this procedure was anticipated to give superior effects than other procedure used in this study
  Other Names: platelet-rich fibrin revascularization
Drug: the effect of apexification in treatment of contaminated and uncontaminated immature permanent teeth — this procedure was anticipated to be replaced by other procedure be used in this study
  Other Names: calcium hydroxide apexification

SUMMARY:
The goal of this clinical trial is to evaluate the effect of platelet-rich fibrin for revascularization of immature permanent teeth in comparison to standard apexification using calcium hydroxide (as a 12 months follow up for previous study) through using clinical outcomes and radiographically using cone beam computed tomography the main questions it aims to answer are

* is the platelet-rich fibrin an effective mean for management of necrotic immature permanent teeth
* is the platelet-rich fibrin has a superior clinical and radiographic effects than calcium hydroxide apexification participants were treated either by platelet-rich fibrin revascularisation or calcium hydroxide apexification

DETAILED DESCRIPTION:
This study is an extension of a previous study [12], encompassing a 12-month fol-low-up period. The protocol for this study received approval from the ethical committee of the Faculty of Dentistry at Mansoura University (11111218) as a randomized con-trolled-clinical trial with a 1:1 allocation ratio for groups and subgroups. The sample size for this study was calculated based on Nagy et al.'s study [13], which determined a re-quired sample size of 28 teeth.

Inclusion and diagnostic criteria:

A total of 28 children, including both boys and girls, were recruited through daily pa-tient screenings in the Clinics of Pediatric Dentistry and dental public health department, Faculty of Dentistry at Mansoura University, following specific inclusion and diagnostic criteria:

* Patients were free of chronic systemic diseases.
* Clinically, a negative response to electric pulp sensibility testing confirmed the pres-ence of immature necrotic permanent teeth.
* Teeth were categorized as uncontaminated if, during the examination, there were no signs of pain, no tenderness during apical percussion, no tenderness of adjacent soft tissues, and no history of open sinus, fistula or swelling.
* Radiographically, teeth were with roots exhibiting thin dentin walls and open apical foramina larger than 1 mm, along with apical periodontitis (considered as contami-nated) or without apical periodontitis (considered as uncontaminated).

Patients' allocation:

The included 28 children were divided into two main groups, each consisting of 14 children: Group I (contaminated teeth) and Group II (uncontaminated teeth). Within each group, children were further divided into two subgroups based on the treatment tech-nique. The allocation was determined through simple randomization, resulting in a Platelet-Rich Fibrin subgroup (n=7 for each) and a Calcium Hydroxide (CH) apexification subgroups (control) (n=7 for each),

ELIGIBILITY:
Inclusion Criteria:

* • Patients were free of chronic systemic diseases.

  * Clinically, a negative response to electric pulp sensibility testing confirmed the pres-ence of immature necrotic permanent teeth.
  * Teeth were categorized as uncontaminated if, during the examination, there were no signs of pain, no tenderness during apical percussion, no tenderness of adjacent soft tissues, and no history of open sinus, fistula or swelling.
  * Radiographically, teeth were with roots exhibiting thin dentin walls and open apical foramina larger than 1 mm, along with apical periodontitis (considered as contami-nated) or without apical periodontitis (considered as uncontaminated).

Exclusion Criteria:

* other than inclusion criteria

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Radiographic measurements of the change in the canal space | 16 months
  Radiographic measurements of the change in the canal space, including an increase in root length and thickness, and reduction in a diameter of the apical foramen, were conducted using the CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Mansoura, Egypt

IPD SHARING:
Plan to Share IPD: No